CLINICAL TRIAL: NCT05804760
Title: Predictive Value of Reduced Keratinized Mucosa on the Secondary Prevention of Peri-implant Mucositis and Periimplantitis in Patients Attending Regular Supportive Peri-implant Care. A Longitudinal Analysis
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 9228_BO_S_2020
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Peri-Implantitis; Peri-implant Mucositis; Lack of Keratinized Gingiva
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- General population (i): All participants of the study, including any periodontal condition.
  Interventions: Diagnostic Test: Measurement of implant parameters
- Periodontally healthy patients with history of periodontitis (ii): Patients whose current periodontal condition is healthy but who have developed periodontitis in the past.
  Interventions: Diagnostic Test: Measurement of implant parameters
- Periodontally healthy patients without history of periodontitis (iii): Patients whose current periodontal condition is healthy, who have also not had periodontitis in the past.
  Interventions: Diagnostic Test: Measurement of implant parameters

INTERVENTIONS:
Diagnostic Test: Measurement of implant parameters — 1. Examination of the inclusion criteria
  2. Medical history/patient-specific data (smoking, tumour diseases, radiation, gender, number of implants, history of periodontitis).
  3. Recording of implant-specific parameters (measurement depth at six sites per implant(probing depth/PD), bleeding and or pus on probing (BOP) at six measurement sites per implant, condition of the peri-implant mucosa using the modified plaque index(mPI) and the modified ginigiva index (mGI), measurement of the width of the keratinised mucosa(KM), type of denture, approximal plaque index (API), radiographically detectable bone resorption.

SUMMARY:
* Capture of the potential risk factor "lack of band of keratinised mucosa" over a period of up to 5 years.
* Recording of peri-implant inflammatory processes in study participants that are not recorded during normal tooth cleaning
* Registration of the extent of radiographic bone loss. Bone resorption through analysis of existing X-ray images
* Individual therapy recommendation/individual supportive peri-implant care in case of peri-implant inflammation
* The present study was specifically designed to investigate the effect of reduced width of keratinized mucosa (KM) on the secondary prevention of peri-implant mucositis and peri-implantitis in patients attending a supportive peri-implant care program (SPIC) over an observation period of up to five years.

DETAILED DESCRIPTION:
Patient information such as age, gender, history of periodontitis, edentulism, previous oral and maxillofacial tumor with a history of head and neck radiation, smoking habits, and metabolic diseases like diabetes mellitus were collected. Implant-specific information such as bone augmentation, year of implantation, implant position, implant level (bone level, tissue level), and number of implants were also documented. Prosthetic factors like the type of prosthesis (single crown, bridge construction, telescope prosthesis) and the type of attachment (cemented, screwed) were recorded. Clinical examination and measurement of clinical parameters were subsequently performed, including probing depth (PD) at six implant sites using a graduated periodontal probe, bleeding on probing or suppuration (BoP/Sup) occurring within 30 seconds after probing, and recessions measured in mm using a graduated periodontal probe between a defined clinical reference point and the implant mucosa.Participants were motivated to undergo regular SPIC, with frequency based on their individual risk factors. Patients without increased risk were encouraged to attend a 6-month recall. If bleeding or suppuration occurred, the frequency of SPIC was increased to monthly controls with oral hygiene instruction and plaque removal. Peri-implantitis therapy was initiated in patients with radiographically detectable bone loss, followed by lifelong SPIC. The modified plaque index (mPl) and full mouth plaque score API were used to assess local plaque accumulation and compliance. The modified gingival index (mGI) was used to assess the inflammatory state of the soft tissue. The mucositis severity score (MSS) was used to investigate the initiation and progression of peri-implant mucositis, with scores ≥18 indicating advanced inflammation. KM impact on MSS values <8 and ≥18 was investigated. Periodontal screening index (PSI) was used to classify the general periodontal condition of the patients by dividing the dentition into sextants. The width of the KM mucogingival junction was assessed using the "rolling technique." Radiographs were analyzed using byzznxt to diagnose possible radiological bone resorption. An individual diagnosis was made for each implant at the end of the examination, and data was collected following a standardized operating procedure and saved electronically.

ELIGIBILITY:
Inclusion Criteria:

- Patients aged at least 18 years who have at least one root-form dental implant in situ and were part of the first (DOI10.1111/clr.13432) and/or the second (DOI 10.1007/s00784-020-03422-1) observational study

Exclusion Criteria:

* Systemic antibiotic use up to 3 months before the examination
* pregnancy
* lactating mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 104 patients with at least one root-shaped dental implant who took part in one of the previous studies and who were attending supportive peri-implant care (SPIC) at the Department of Prosthetic Dentistry and Biomedical Materials Science of Hannover Medical School were asked to participate in the study.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Protective value of keratinized mucosa around dental implants in periodontal healthy patients | Up to five years
  Keratinized mucosa is a significant protective factor for the progression of peri-implant mucositis to severe peri-implant mucositis and to peri-implantitis in patients without history of periodontitis attending regular SPIC over a period of up to five years.

SECONDARY OUTCOMES:
Mucositis severity score (MSS) related to the supported peri implant care (SPIC) | Up to five years
  1. The MSS ≤6 is a reasonable cut-off to define the endpoint of peri-implantitis treatment, define the entrance of the patient into SPIC and is an indicator for a successful SPIC program.
  2. MSS scores 7-17 indicate an elevated risk of disease progression and support the clinicians in decision making on reevaluating frequency and protocol of the patients individual SPIC.
  3. MSS scores ≥18 indicate that SPIC is not enough and (non-) surgical peri-implantitis treatment should be considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Hochschule Hannover (MHH), Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided